CLINICAL TRIAL: NCT07171567
Title: Vacuum Therapy for the Treatment of Penile Numbness/Sensory Changes
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 20250231-01H
Record Dates: First submitted 2025-08-26; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Penile Numbness
Keywords: Penile numbness; Penile sensation changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- vacuum erection device (VED) (Experimental)
  Interventions: Device: Vacuum erection device

INTERVENTIONS:
Device: Vacuum erection device — A vacuum erection device (VED) is a mechanical device designed to enhance blood flow to the corpora cavernosa by creating a vacuum environment. When combined with a constriction ring at the base of the penis, VEDs can promote and sustain an erection.
  This is a prospective, uncontrolled, hypothesis-generating pilot study. Eight adult male participants with penile insensitivity will be enrolled and asked to use a VED daily for six months. Monthly self-reported questionnaire data and biweekly follow-up calls will be used to assess feasibility and to collect exploratory outcome data.

SUMMARY:
This is a prospective, uncontrolled, Hypothesis generating study. A total of eight adult male participants experiencing penile insensitivity will be recruited through the Ottawa Hospital's Men's Health Clinic. Participants will receive a Health Canada Class I VED to use daily over a six-month period. The study includes biweekly check-ins and monthly questionnaire assessments (including the IIEF-5 and two custom instruments focused on penile sensitivity) administered via Lime Survey.

The primary outcome is to explore the feasibility and acceptability of daily vacuum erection device (VED) therapy over a 6-month period in adult males experiencing penile numbness/insensitivity. Data analysis will focus on feasibility metrics (e.g., adherence rates, completion of assessments) and descriptive statistics. Any changes in questionnaire scores over time will be evaluated using within-subject comparisons (e.g., Wilcoxon signed-rank test), recognizing that findings are preliminary and not generalizable due to the lack of a control group.

ELIGIBILITY:
Inclusion Criteria

* Male adults (age 18 and over)
* Have been seen by a urologist in consultation for penile numbness/insensitivity

5.2 Exclusion Criteria

- Under 18 years of age

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment to study | 6 months
  To evaluate the feasibility of recruitment to a study examining the daily use of vacuum erection device (VED) therapy over a 6-month period in adult males with penile numbness or reduced sensation. Feasibility will be assessed via the ability to enroll subjects within a 1 year period and by treatment adherence and completion rates. Treatment adherence/completion will be assessed during standardized study visits
Acceptability of treatment | 6 months
  Acceptability will be evaluated through patient-reported experiences using online questionnaires. Changes in penile sensation will be measured using patient-reported outcomes of erectile function (standardized questionnaires) and a subjective Likert scale of penile numbness collected at baseline, throughout the study and at the end of the 6-month intervention

CONTACTS AND LOCATIONS:
Overall Officials: Luke Witherspoon, Principal Investigator — The Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No